CLINICAL TRIAL: NCT02084017
Title: Single Center Prospective Randomized Control Trial on Negative Pressure Wound Therapy for Primarily Closed Groin Incisions Following Lower-limb Re-vascularization to Reduce Surgical Site Infection
Brief Title: Negative Pressure Wound Therapy for the Prevention of Surgical Site Infection Following Lower Limb Revascularization
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Adam Power, Principle Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RRG-104871
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Surgical Wound Infection; Peripheral Vascular Diseases
Keywords: Surgical Site Infection; Vascular Surgery; Negative Pressure Wound Therapy
MeSH Terms: conditions — Surgical Wound Infection; Peripheral Vascular Diseases | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current Standard (Active Comparator): Standard Tegaderm (3M Healthcare, St. Paul, MN) adhesive dressing applied under sterile conditions in the operating room following skin closure. Dressing changed post-operative day two and daily thereafter with daily inspection for infection by a physician.
  Interventions: Device: Standard Tegaderm (3M Healthcare, St. Paul, MN) adhesive dressing
- Negative Pressure Wound Therapy (Experimental): A negative pressure therapy (Kinetic Concepts, Inc, San Antionio, Tex) device will be applied under sterile conditions post-operatively and placed on suction (125-150 cm H2O). The device will be removed on post-operative day 4-7 depending on day of discharge.
  Interventions: Device: Prevena (Negative Pressure Wound Therapy Device)

INTERVENTIONS:
Device: Prevena (Negative Pressure Wound Therapy Device) — No other details required.
  Other Names: Prevena; Prevena Incision Management System; Negative Pressure Wound Therapy Device; Vacuum Therapy
  Arms: Negative Pressure Wound Therapy
Device: Standard Tegaderm (3M Healthcare, St. Paul, MN) adhesive dressing
  Arms: Current Standard

SUMMARY:
The purpose of this study is to investigate the current standard of wound care following vascular operations compared to to a negative pressure wound therapy (vacuum dressing) and the rate of surgical site infections (SSIs) in patients undergoing surgery to restore blood flow to the lower limb(s).

Negative pressure wound therapy consists of a closed, sealed system that produces negative pressure (vacuum) to the wound surface. The device itself consists of open-cell foam that is sealed with an occlusive adhesive dressing (covers and sticks to the incision) and suction is maintained by connecting suction tubes to a vacuum pump and waste collector.

The investigators objectives are to determine whether there will be any reduction in surgical site infection and this potential reduction will influence length of hospital stay, emergency room visits, antibiotic use and need for re-operation.

DETAILED DESCRIPTION:
The study is a non-blinded randomized control trial. The study examines the effect on wound healing and surgical site infection using negative pressure wound therapy compared to standard dressing in high-risk patients (BMI > 30, previous femoral cut-down). The investigators expected to find a lower surgical site infection rate in patients using the NPWT device.

Patients after giving informed consent will be randomized to receive either NPWT or standard wound therapy following tier lower-limb revascularization operative. Both will be applied under sterile conditions immediately post-operatively. The intervention will be left for 4-7 days depending on the discharge date and the standard dressing will be removed on post-operative day two.

The data will be analyzed with an intention to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* Previous femoral exposure
* Undergoing lower-limb revascularization

Exclusion Criteria:

* Cannot obtain seal
* Non-primary wound closure
* Pre-existing infection
* Endovascular repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-10 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 30 days
  Surgical site infection is defined by the CDC Guidelines for surgical site infection and by the Szilagyi classification of vascular wound infections.

SECONDARY OUTCOMES:
Length of stay | Date of discharge
  Duration (in days) the patient stays in hospital post-operatively
Emergency room visits | 30 days
  Number of times the patient return to the emergency department following discharge from hospital and before the follow-up clinic appointment
All-cause mortality | 30 days
Re-operation rate | 30 days
  Need for re-operation following graft failure secondary to infection
Amputation | 30 days
  Need for amputation post-operatively secondary to infection

CONTACTS AND LOCATIONS:
Overall Officials: Adam Power, MD, Principal Investigator — London Health Sciences Center
Locations (1):
- Victoria Hospital, London, Ontario, Canada

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835
- [Derived] Lee K, Murphy PB, Ingves MV, Duncan A, DeRose G, Dubois L, Forbes TL, Power A. Randomized clinical trial of negative pressure wound therapy for high-risk groin wounds in lower extremity revascularization. J Vasc Surg. 2017 Dec;66(6):1814-1819. doi: 10.1016/j.jvs.2017.06.084. Epub 2017 Aug 31. PMID 28865981
- [Derived] Murphy P, Lee K, Dubois L, DeRose G, Forbes T, Power A. Negative pressure wound therapy for high-risk wounds in lower extremity revascularization: study protocol for a randomized controlled trial. Trials. 2015 Nov 4;16:504. doi: 10.1186/s13063-015-1026-1. PMID 26537879